CLINICAL TRIAL: NCT03203486
Title: The Effectiveness of a Mediterranean Diet Intervention in NAFLD Clinical Course
Brief Title: Response of NAFLD Patients to Mediterranean Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: National and Kapodistrian University of Athens (Other); Greek Secretariat for Research and Technology (Unknown)
Responsible Party: Principal Investigator, Andriana C Kaliora, Assistant Professor, Human Nutrition and Foods, Harokopio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 09-ΣΥΝ-12-890
Record Dates: First submitted 2017-06-26; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: NAFLD; Steatosis of Liver
Keywords: NAFLD; no fibrosis; Mediterranean diet; STAT3; GCKR; visfatin; oxidized LDL; fasting glucose; inflammation
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Inflammation | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: non-randomised, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meditteranean Diet (Experimental): NAFLD patients attended appointments with experienced dieticians to receive nutritional guidance based on a traditional Mediterranean Diet for 6 months.
  Interventions: Other: Mediterranean Diet

INTERVENTIONS:
Other: Mediterranean Diet — Participants were instructed to include vegetables, whole grains and fruits in their diet and increase fish, legumes and raw nut intake. Emphasis was given to extra virgin olive oil as the main added fat in meals. Particular attention was drained to decrease fermented dairy and poultry, with small amounts of red meat and homemade sweets. All participants were given meal plans in which the distribution of nutrients in relation to total caloric value was as follows: 40% of total energy as fat (50% as MUFAs), 20% as protein, 40% as carbohydrate, 300mg/d as dietary cholesterol and 20-30g fiber/d.

SUMMARY:
The effects of Mediterranean Diet (MedDiet) on clinical, biochemical and inflammatory profile in NAFLD patients with simple steatosis. Potential associations of single nucleotide polymorphisms to diet composition and patients' profile were also investigated.

DETAILED DESCRIPTION:
Diet is a modifiable key factor targeted in prevention and management of non-alcoholic fatty liver disease (NAFLD). The aim of the study is to investigate the effect of Mediterranean Diet (MedDiet) on clinical, biochemical and inflammatory profile in NAFLD patients with simple steatosis. Potential associations of single nucleotide polymorphisms to diet composition and patients' profile are investigated. In this non-randomised, open-label study, 44 untreated NAFLD patients with non significant fibrosis receive nutritional counsel to increase adherence to MedDiet. Adherence to MedDiet is estimated with MedDietScore. Furthermore, genotyping of STAT3 rs2293152 and GCKR rs1260326 single nucleotide polymorphisms takes place.

ELIGIBILITY:
Inclusion Criteria:

* men and women >18y of age, no change in body weight (BW) for the last 6 months prior to the trial and body mass index (BMI) >25 kg/m2.

Exclusion Criteria:

* the presence of chronic viral hepatitis, the presence of congenital or acquired liver disease, the history of prior exposure to hepatotoxic drugs, the evidence of hepatic cirrhosis, ultrasonography values less than 1Hz, bariatric surgery, daily consumption of ethanol more than 20g for women and more than 30g for men for over 6 months during the last 5 years, any medication effective on fatty liver disease introduced <6 months prior to or during the trial, the co-presence of a life-threatening disease, psychiatric disorders impairing the patient's ability to provide written informed consent, age>65 years, pregnant or lactating women, subjects supplemented with omega-3 polyunsaturated fatty acids, probiotics/synbiotics, antioxidant vitamins and/or phytochemicals, any planned, structured and repetitive physical activity. Patients with any medication change during the trial were excluded from analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Regulation of hepatic steatosis | Change from Baseline to 6 months
  A decrease in liver fat

SECONDARY OUTCOMES:
Adherence to MedDiet | Change from Baseline to 6 months
  Increase in MedDietScore
Regulation of visfatin | Change from Baseline to 6 months
  Decrease in visfatin levels
Regulation of oxLDL | Change from Baseline to 6 months
  Decrease in oxLDL levels
Association of single nucleotide polymorphisms to response to dietary treatment | Change from Baseline to 6 months
  Decrease in visfatin in carriers of the risk allele

CONTACTS AND LOCATIONS:
Overall Officials: Andriana C Kaliora, PhD, Principal Investigator — Harokopio University of Athens

IPD SHARING:
Plan to Share IPD: No